CLINICAL TRIAL: NCT06030115
Title: Effects of a Physical Therapist-driven Individualized Hybrid Model of the Exercise Component of Cardiac Rehabilitation on Patient Outcomes: a Prospective Cohort Study
Brief Title: Effects of a Hybrid Model of Cardiac Rehabilitation on Patient Outcomes
Status: Completed | Type: Observational
Sponsor: Good Shepherd Integrated Healthcare Systems (Other)
Responsible Party: Principal Investigator, Kevin Minchin, Physical Therapist, Rehabilitation Director, Good Shepherd Integrated Healthcare Systems
Other Study IDs: GoodShepherdIHS
Record Dates: First submitted 2023-08-24; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Graft CABG; Stent; Valve Replacement
Keywords: Physical Therapy; Cardiopulmonary Rehabilitation; Cardiac Surgery; Exercise; Heart Rate; Objective Outcome Assessments
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Rehab Patients: All participants referred to the clinic meeting the inclusion and exclusion criteria who wanted to participate in the study.
  Interventions: Other: Exercise Component Of Cardiac Rehabilitation (Hybrid Model) Intensity Recovery Progression Protocol (IRPP)

INTERVENTIONS:
Other: Exercise Component Of Cardiac Rehabilitation (Hybrid Model) Intensity Recovery Progression Protocol (IRPP) — Data collected on participants who completed the intensity recovery progression protocol program

SUMMARY:
Determine if the standard of care at a cardiac rehabilitation center using what the investigators term to be "hybrid model" on the exercise component of cardiac rehabilitation is associated with improved adherence and outcomes. Discuss the hybrid model in comparison to traditional cardiac rehabilitation and layout a template on how to incorporate this hybrid model. Discuss factors that may lead to poor adherence and attendance to cardiac rehabilitation.

DETAILED DESCRIPTION:
Purpose: The aim of this prospective cohort study was to determine the effectiveness of an individualized physical therapist (PT) driven hybrid model of the exercise component of cardiac rehabilitation (CR) that uses a novel intensity-recovery progression protocol (IRPP) and cardiac testing template (CTT) to assess achieved heart rate intensity (AHRI%), heart rate recovery (HRR%), and intensity-recovery total (IR%) as indicators to guide treatment.

Methods: Assessment of a subjective questionnaire, vital signs, treadmill 6-minute walk (6MW), 1-minute sit-to-stand (1STS), 1-minute step (1ST), and 1-minute agility square tests (1AST) were assessed on 100 participants during the 36-visit program. The hybrid model was led by a PT, was longer in duration, added high intensity interval training (HIIT) to continuous aerobic exercise training (CAET) and resistance training, and used a 1:1 treatment ratio. Treatment intensity and progression were measured based on clinical decision making through the IRPP and CTT.

ELIGIBILITY:
Inclusion Criteria:

* Underwent cardiac surgery (CABG, PCI with stent placement, and valve replacement)
* Surgery was within the previous 365 days
* Could independently ambulate into the facility.

Exclusion Criteria:

* Implantable cardioverter defibrillator (ICD)
* Pacemaker (PPM)
* Heart Transplant
* Left ventricular assist device (LVAD)
* All other cardiac procedures not listed within inclusion criteria
* Diagnosed a-fib
* Participants who attended cardiac rehabilitation before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants analyzed (73 males, 27 females) had an average starting age of 66.1 years (SD=9.6; range 41-88 years). The admitting diagnoses were 50% stent, 37% CABG, 8% valve replacement and 5% a combination of the above.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | Six Minutes
  Treadmill Six Minute Walk Test
Timed Sit To Stand Test | One Minute
  A standardized test measuring how many times an individual can stand from a standardized seated position in one minute using hand support to push off.
Timed Step Test | One Minute
  A test measuring how many repetitions an individual can go up and down a standardized step while using bilateral arm support on a rail.
Timed Agility Square Test | One Minute
  Using agility ladder square to go in and out of designated two boxes
Achieved Target Heart Rate (AHRI%) | One minute
  Heart rate achieved during outcome measurements (six minute walk test, timed sit to stand test, timed step test, timed agility square test). Completed every 5 visits from date of initiation up to 1 year after initiation or until visit 36 achieved (whichever comes first). Participants expected to attend the program at a frequency of 2x a week for 36 total visits.
Heart Rate Recovery (HRR%) | One minute
  Heart rate observed one minute after outcome measurements (six minute walk test, timed sit to stand test, timed step test, timed agility square test). Completed every 5 visits from date of initiation up to 1 year after initiation or until visit 36 achieved (whichever comes first).
Intensity Recovery Total Score (IR%) | One minute
  The total of the AHRI + HRR during objective measurements (six minute walk test, timed sit to stand test, timed step test, timed agility square test). Completed every 5 visits from date of initiation up to 1 year after initiation or until visit 36 achieved (whichever comes first).
Subjective Questionnaire | From date of initiation of study up to 1 year after initiation. Collected on Visit 1, Visit 15, Visit 30 for each participant, who were expected to attend the program at a frequency of 2x a week for 36 total sessions.
  Three questions (where higher scores denote better outcomes) Question 1: Rate your endurance (using a visual analog scale from 0-100% marked every 10%)? Question 2: Estimate how many stairs you could go up using arm support before you would have to take a break? Question 3: Estimate how many hours of exercise you completed in the previous 7 days?

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Minchin, DPT, Principal Investigator — Good Shepherd
Locations (1):
- Good Shepherd Integrated Healthcare Systems, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
IPD (decodified) will be stored in a password protected laptop in a locked room in a locked file cabinet at the clinic site. The statistical summarized analysis will be the main focus for the public and other researchers. The cardiac testing template in excel format will be available for other researchers looking to use the hybrid model explained in the study, however, this template will not contain individualized personal data.

REFERENCES:
- [Background] National Vital Statistics System. Mortality Mulitple Cause-of-Death: Centers for Disease Control adn Prevention; 2021 [Available from:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; Society of Cardiovascular Anesthesiologists; Society of Thoracic Surgeons. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Developed in collaboration with the American Association for Thoracic Surgery, Society of Cardiovascular Anesthesiologists, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2011 Dec 6;58(24):e123-210. doi: 10.1016/j.jacc.2011.08.009. Epub 2011 Nov 7. No abstract available. PMID 22070836
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; ACCF; AHA; SCAI. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2012 Feb 15;79(3):453-95. doi: 10.1002/ccd.23438. No abstract available. PMID 22328235
- [Background] Wenger NK. Current status of cardiac rehabilitation. J Am Coll Cardiol. 2008 Apr 29;51(17):1619-31. doi: 10.1016/j.jacc.2008.01.030. PMID 18436113
- [Background] Winzer EB, Woitek F, Linke A. Physical Activity in the Prevention and Treatment of Coronary Artery Disease. J Am Heart Assoc. 2018 Feb 8;7(4):e007725. doi: 10.1161/JAHA.117.007725. No abstract available. PMID 29437600
- [Background] Origuchi H, Itoh H, Momomura SI, Nohara R, Daida H, Masuda T, Kohzuki M, Makita S, Ueshima K, Nagayama M, Omiya K, Adachi H, Goto Y. Active Participation in Outpatient Cardiac Rehabilitation Is Associated With Better Prognosis After Coronary Artery Bypass Graft Surgery - J-REHAB CABG Study. Circ J. 2020 Feb 25;84(3):427-435. doi: 10.1253/circj.CJ-19-0650. Epub 2020 Feb 8. PMID 32037378
- [Background] Mampuya WM. Cardiac rehabilitation past, present and future: an overview. Cardiovasc Diagn Ther. 2012 Mar;2(1):38-49. doi: 10.3978/j.issn.2223-3652.2012.01.02. PMID 24282695
- [Background] Keteyian SJ, Jackson SL, Chang A, Brawner CA, Wall HK, Forman DE, Sukul D, Ritchey MD, Sperling LS. Tracking Cardiac Rehabilitation Utilization in Medicare Beneficiaries: 2017 UPDATE. J Cardiopulm Rehabil Prev. 2022 Jul 1;42(4):235-245. doi: 10.1097/HCR.0000000000000675. Epub 2022 Feb 8. PMID 35135961
- [Background] Ritchey MD, Maresh S, McNeely J, Shaffer T, Jackson SL, Keteyian SJ, Brawner CA, Whooley MA, Chang T, Stolp H, Schieb L, Wright J. Tracking Cardiac Rehabilitation Participation and Completion Among Medicare Beneficiaries to Inform the Efforts of a National Initiative. Circ Cardiovasc Qual Outcomes. 2020 Jan;13(1):e005902. doi: 10.1161/CIRCOUTCOMES.119.005902. Epub 2020 Jan 14. PMID 31931615
- [Background] Thomas RJ, Balady G, Banka G, Beckie TM, Chiu J, Gokak S, Ho PM, Keteyian SJ, King M, Lui K, Pack Q, Sanderson BK, Wang TY. 2018 ACC/AHA Clinical Performance and Quality Measures for Cardiac Rehabilitation: A Report of the American College of Cardiology/American Heart Association Task Force on Performance Measures. J Am Coll Cardiol. 2018 Apr 24;71(16):1814-1837. doi: 10.1016/j.jacc.2018.01.004. Epub 2018 Mar 29. No abstract available. PMID 29606402
- [Background] Beatty AL, Li S, Thomas L, Amsterdam EA, Alexander KP, Whooley MA. Trends in referral to cardiac rehabilitation after myocardial infarction: data from the National Cardiovascular Data Registry 2007 to 2012. J Am Coll Cardiol. 2014 Jun 17;63(23):2582-2583. doi: 10.1016/j.jacc.2014.03.030. Epub 2014 Apr 23. No abstract available. PMID 24768872
- [Background] Peters AE, Keeley EC. Trends and Predictors of Participation in Cardiac Rehabilitation Following Acute Myocardial Infarction: Data From the Behavioral Risk Factor Surveillance System. J Am Heart Assoc. 2017 Dec 29;7(1):e007664. doi: 10.1161/JAHA.117.007664. PMID 29288154
- [Background] Resurreccion DM, Motrico E, Rigabert A, Rubio-Valera M, Conejo-Ceron S, Pastor L, Moreno-Peral P. Barriers for Nonparticipation and Dropout of Women in Cardiac Rehabilitation Programs: A Systematic Review. J Womens Health (Larchmt). 2017 Aug;26(8):849-859. doi: 10.1089/jwh.2016.6249. Epub 2017 Apr 7. PMID 28388314
- [Background] Lee M, Wood T, Chan S, Marziali E, Tang T, Banner D, Lear SA. Cardiac rehabilitation program: An exploration of patient experiences and perspectives on program dropout. Worldviews Evid Based Nurs. 2022 Feb;19(1):56-63. doi: 10.1111/wvn.12554. Epub 2022 Jan 17. PMID 35040245
- [Background] Squires RW, Kaminsky LA, Porcari JP, Ruff JE, Savage PD, Williams MA. Progression of Exercise Training in Early Outpatient Cardiac Rehabilitation: AN OFFICIAL STATEMENT FROM THE AMERICAN ASSOCIATION OF CARDIOVASCULAR AND PULMONARY REHABILITATION. J Cardiopulm Rehabil Prev. 2018 May;38(3):139-146. doi: 10.1097/HCR.0000000000000337. PMID 29697494
- [Background] Franklin B, Fern A, Fowler A, Spring T, Dejong A. Exercise physiologist's role in clinical practice. Br J Sports Med. 2009 Feb;43(2):93-8. doi: 10.1136/bjsm.2008.055202. Epub 2008 Dec 2. PMID 19050005
- [Background] Balady GJ, Williams MA, Ades PA, Bittner V, Comoss P, Foody JA, Franklin B, Sanderson B, Southard D; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee; Council on Clinical Cardiology; Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; American Association of Cardiovascular and Pulmonary Rehabilitation. Core components of cardiac rehabilitation/secondary prevention programs: 2007 update: a scientific statement from the American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; the Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; and the American Association of Cardiovascular and Pulmonary Rehabilitation. J Cardiopulm Rehabil Prev. 2007 May-Jun;27(3):121-9. doi: 10.1097/01.HCR.0000270696.01635.aa. PMID 17558191
- [Background] Williams MA, Haskell WL, Ades PA, Amsterdam EA, Bittner V, Franklin BA, Gulanick M, Laing ST, Stewart KJ; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Nutrition, Physical Activity, and Metabolism. Resistance exercise in individuals with and without cardiovascular disease: 2007 update: a scientific statement from the American Heart Association Council on Clinical Cardiology and Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2007 Jul 31;116(5):572-84. doi: 10.1161/CIRCULATIONAHA.107.185214. Epub 2007 Jul 16. PMID 17638929
- [Background] Price KJ, Gordon BA, Bird SR, Benson AC. A review of guidelines for cardiac rehabilitation exercise programmes: Is there an international consensus? Eur J Prev Cardiol. 2016 Nov;23(16):1715-1733. doi: 10.1177/2047487316657669. Epub 2016 Jun 27. PMID 27353128
- [Background] Villelabeitia-Jaureguizar K, Vicente-Campos D, Senen AB, Jimenez VH, Garrido-Lestache MEB, Chicharro JL. Effects of high-intensity interval versus continuous exercise training on post-exercise heart rate recovery in coronary heart-disease patients. Int J Cardiol. 2017 Oct 1;244:17-23. doi: 10.1016/j.ijcard.2017.06.067. Epub 2017 Jun 17. PMID 28648356
- [Background] Wehmeier UF, Schweitzer A, Jansen A, Probst H, Gruter S, Hahnchen S, Hilberg T. Effects of high-intensity interval training in a three-week cardiovascular rehabilitation: a randomized controlled trial. Clin Rehabil. 2020 May;34(5):646-655. doi: 10.1177/0269215520912302. Epub 2020 Mar 16. PMID 32172602
- [Background] Papathanasiou JV, Petrov I, Tokmakova MP, Dimitrova DD, Spasov L, Dzhafer NS, Tsekoura D, Dionyssiotis Y, Ferreira AS, Lopes AJ, Rosulescu E, Foti C. Group-based cardiac rehabilitation interventions. A challenge for physical and rehabilitation medicine physicians: a randomized controlled trial. Eur J Phys Rehabil Med. 2020 Aug;56(4):479-488. doi: 10.23736/S1973-9087.20.06013-X. Epub 2020 Jan 23. PMID 31976639
- [Background] Dun Y, Smith JR, Liu S, Olson TP. High-Intensity Interval Training in Cardiac Rehabilitation. Clin Geriatr Med. 2019 Nov;35(4):469-487. doi: 10.1016/j.cger.2019.07.011. Epub 2019 Jul 12. PMID 31543179
- [Background] Shah BR, Cowper PA, O'Brien SM, Jensen N, Drawz M, Patel MR, Douglas PS, Peterson ED. Patterns of cardiac stress testing after revascularization in community practice. J Am Coll Cardiol. 2010 Oct 12;56(16):1328-34. doi: 10.1016/j.jacc.2010.03.093. PMID 20888523
- [Background] Noonan V, Dean E. Submaximal exercise testing: clinical application and interpretation. Phys Ther. 2000 Aug;80(8):782-807. PMID 10911416
- [Background] Dean E, Lomi C. A health and lifestyle framework: An evidence-informed basis for contemporary physical therapist clinical practice guidelines with special reference to individuals with heart failure. Physiother Res Int. 2022 Jul;27(3):e1950. doi: 10.1002/pri.1950. Epub 2022 Apr 25. PMID 35467065
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] KARVONEN MJ, KENTALA E, MUSTALA O. The effects of training on heart rate; a longitudinal study. Ann Med Exp Biol Fenn. 1957;35(3):307-15. No abstract available. PMID 13470504
- [Background] Facioli TP, Philbois SV, Gastaldi AC, Almeida DS, Maida KD, Rodrigues JAL, Sanchez-Delgado JC, Souza HCD. Study of heart rate recovery and cardiovascular autonomic modulation in healthy participants after submaximal exercise. Sci Rep. 2021 Feb 11;11(1):3620. doi: 10.1038/s41598-021-83071-w. PMID 33574441
- [Background] American College of Sports Medicine, Riebe D, Ehrman JK, Liguori G, Magal M. ACSM's guidelines for exercise testing and prescription. Tenth edition. ed. Philadelphia: Wolters Kluwer; 2018. xxx, 472 pages p.
- [Background] Stevens D, Elpern E, Sharma K, Szidon P, Ankin M, Kesten S. Comparison of hallway and treadmill six-minute walk tests. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1540-3. doi: 10.1164/ajrccm.160.5.9808139. PMID 10556117
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Lenssen AF, Wijnen LC, Vankan DG, Van Eck BH, Berghmans DP, Roox GM. Six-minute walking test done in a hallway or on a treadmill: how close do the two methods agree? Eur J Cardiovasc Prev Rehabil. 2010 Dec;17(6):713-7. doi: 10.1097/HJR.0b013e32833a1963. PMID 20431392
- [Background] Fyderyk Prochaczek JSB, Witold Żmuda, Katarzyna R. Świda, Zbigniew W. Szczurek, Jerzy, Winiarska GaA. The Six-Minute Walk Test on the Treadmill, Chronic Obstructive Pulmonary Disease - Current Concepts and Practice. Ong DK-C, editor: InTech; 2012.
- [Background] Gochicoa-Rangel L, Ramirez-Jose MC, Troncoso-Huitron P, Silva-Ceron M, Guzman-Valderrabano C, Lechuga-Trejo I, Cid-Juarez S, Torre-Bouscoulet L. Shorter corridors can be used for the six-minute walk test in subjects with chronic lung diseases. Respir Investig. 2020 Jul;58(4):255-261. doi: 10.1016/j.resinv.2019.12.009. Epub 2020 Feb 26. PMID 32111517
- [Background] Scivoletto G, Tamburella F, Laurenza L, Foti C, Ditunno JF, Molinari M. Validity and reliability of the 10-m walk test and the 6-min walk test in spinal cord injury patients. Spinal Cord. 2011 Jun;49(6):736-40. doi: 10.1038/sc.2010.180. Epub 2011 Jan 11. PMID 21221120
- [Background] de Almeida FG, Victor EG, Rizzo JA. Hallway versus treadmill 6-minute-walk tests in patients with chronic obstructive pulmonary disease. Respir Care. 2009 Dec;54(12):1712-6. PMID 19961638
- [Background] Laskin JJ, Bundy S, Marron H, Moore H, Swanson M, Blair M, Humphrey R. Using a treadmill for the 6-minute walk test: reliability and validity. J Cardiopulm Rehabil Prev. 2007 Nov-Dec;27(6):407-10. doi: 10.1097/01.HCR.0000300270.45881.d0. PMID 18197077
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Crook S, Busching G, Schultz K, Lehbert N, Jelusic D, Keusch S, Wittmann M, Schuler M, Radtke T, Frey M, Turk A, Puhan MA, Frei A. A multicentre validation of the 1-min sit-to-stand test in patients with COPD. Eur Respir J. 2017 Mar 2;49(3):1601871. doi: 10.1183/13993003.01871-2016. Print 2017 Mar. PMID 28254766
- [Background] Christle JW, Schlumberger A, Haller B, Gloeckl R, Halle M, Pressler A. Individualized vs. group exercise in improving quality of life and physical activity in patients with cardiac disease and low exercise capacity: results from the DOPPELHERZ trial. Disabil Rehabil. 2017 Dec;39(25):2566-2571. doi: 10.1080/09638288.2016.1242174. Epub 2016 Oct 28. PMID 27793077
- [Background] Grundtvig M, Eriksen-Volnes T, Orn S, Slind EK, Gullestad L. 6 min walk test is a strong independent predictor of death in outpatients with heart failure. ESC Heart Fail. 2020 Oct;7(5):2904-2911. doi: 10.1002/ehf2.12900. Epub 2020 Jul 17. PMID 32677748
- [Background] Cole CR, Blackstone EH, Pashkow FJ, Snader CE, Lauer MS. Heart-rate recovery immediately after exercise as a predictor of mortality. N Engl J Med. 1999 Oct 28;341(18):1351-7. doi: 10.1056/NEJM199910283411804. PMID 10536127
- [Background] Ghaffari S, Kazemi B, Aliakbarzadeh P. Abnormal heart rate recovery after exercise predicts coronary artery disease severity. Cardiol J. 2011;18(1):47-54. PMID 21305485
- [Background] Lipinski MJ, Vetrovec GW, Gorelik D, Froelicher VF. The importance of heart rate recovery in patients with heart failure or left ventricular systolic dysfunction. J Card Fail. 2005 Oct;11(8):624-30. doi: 10.1016/j.cardfail.2005.06.429. PMID 16230267
- [Background] Sydo N, Sydo T, Gonzalez Carta KA, Hussain N, Farooq S, Murphy JG, Merkely B, Lopez-Jimenez F, Allison TG. Prognostic Performance of Heart Rate Recovery on an Exercise Test in a Primary Prevention Population. J Am Heart Assoc. 2018 Mar 26;7(7):e008143. doi: 10.1161/JAHA.117.008143. PMID 29581219
- [Background] Pierdomenico SD, Bucci A, Lapenna D, Cuccurullo F, Mezzetti A. Heart rate in hypertensive patients treated with ACE inhibitors and long-acting dihydropyridine calcium antagonists. J Cardiovasc Pharmacol. 2002 Aug;40(2):288-95. doi: 10.1097/00005344-200208000-00014. PMID 12131558
- [Background] Paolillo S, Dell'Aversana S, Esposito I, Poccia A, Perrone Filardi P. The use of beta-blockers in patients with heart failure and comorbidities: Doubts, certainties and unsolved issues. Eur J Intern Med. 2021 Jun;88:9-14. doi: 10.1016/j.ejim.2021.03.035. Epub 2021 Apr 30. PMID 33941435
- [Background] White P. Calcium channel blockers. AACN Clin Issues Crit Care Nurs. 1992 May;3(2):437-46. doi: 10.4037/15597768-1992-2015. PMID 1315559
- [Background] Erdmann E. Digitalis therapy--relevance of heart rate reduction. Basic Res Cardiol. 1998;93 Suppl 1:156-9. doi: 10.1007/s003950050244. PMID 9833144
- [Background] Godlasky E, Hoffman T, Weber-Peters S, Bradford R, Miller N, Kunselman AR, Lott MEJ. Effects of beta-Blockers on Maximal Heart Rate Prediction Equations in a Cardiac Population. J Cardiopulm Rehabil Prev. 2018 Mar;38(2):111-117. doi: 10.1097/HCR.0000000000000328. PMID 29465497
- [Background] Harada ND, Chiu V, Stewart AL. Mobility-related function in older adults: assessment with a 6-minute walk test. Arch Phys Med Rehabil. 1999 Jul;80(7):837-41. doi: 10.1016/s0003-9993(99)90236-8. PMID 10414771
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Hamilton DM, Haennel RG. Validity and reliability of the 6-minute walk test in a cardiac rehabilitation population. J Cardiopulm Rehabil. 2000 May-Jun;20(3):156-64. doi: 10.1097/00008483-200005000-00003. PMID 10860197
- [Background] Demers C, McKelvie RS, Negassa A, Yusuf S; RESOLVD Pilot Study Investigators. Reliability, validity, and responsiveness of the six-minute walk test in patients with heart failure. Am Heart J. 2001 Oct;142(4):698-703. doi: 10.1067/mhj.2001.118468. PMID 11579362
- [Background] Bellet RN, Adams L, Morris NR. The 6-minute walk test in outpatient cardiac rehabilitation: validity, reliability and responsiveness--a systematic review. Physiotherapy. 2012 Dec;98(4):277-86. doi: 10.1016/j.physio.2011.11.003. Epub 2012 May 16. PMID 23122432
- [Background] Uszko-Lencer NHMK, Mesquita R, Janssen E, Werter C, Brunner-La Rocca HP, Pitta F, Wouters EFM, Spruit MA. Reliability, construct validity and determinants of 6-minute walk test performance in patients with chronic heart failure. Int J Cardiol. 2017 Aug 1;240:285-290. doi: 10.1016/j.ijcard.2017.02.109. Epub 2017 Feb 28. PMID 28377186
- [Background] Lee MC. Validity of the 6-minute walk test and step test for evaluation of cardio respiratory fitness in patients with type 2 diabetes mellitus. J Exerc Nutrition Biochem. 2018 Mar 30;22(1):49-55. doi: 10.20463/jenb.2018.0008. PMID 29673246
- [Background] Saba MA, Goharpey S, Attarbashi Moghadam B, Salehi R, Nejatian M. Correlation Between the 6-Min Walk Test and Exercise Tolerance Test in Cardiac Rehabilitation After Coronary Artery Bypass Grafting: A Cross-sectional Study. Cardiol Ther. 2021 Jun;10(1):201-209. doi: 10.1007/s40119-021-00210-0. Epub 2021 Feb 13. PMID 33586086
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Tremblay Labrecque PF, Harvey J, Nadreau E, Maltais F, Dion G, Saey D. Validation and Cardiorespiratory Response of the 1-Min Sit-to-Stand Test in Interstitial Lung Disease. Med Sci Sports Exerc. 2020 Dec;52(12):2508-2514. doi: 10.1249/MSS.0000000000002423. PMID 32555023
- [Background] Bohannon RW, Crouch R. 1-Minute Sit-to-Stand Test: SYSTEMATIC REVIEW OF PROCEDURES, PERFORMANCE, AND CLINIMETRIC PROPERTIES. J Cardiopulm Rehabil Prev. 2019 Jan;39(1):2-8. doi: 10.1097/HCR.0000000000000336. PMID 30489442
- [Background] Wang Z, Yan J, Meng S, Li J, Yu Y, Zhang T, Tsang RCC, El-Ansary D, Han J, Jones AYM. Reliability and validity of sit-to-stand test protocols in patients with coronary artery disease. Front Cardiovasc Med. 2022 Aug 25;9:841453. doi: 10.3389/fcvm.2022.841453. eCollection 2022. PMID 36093135
- [Background] Kohlbrenner D, Benden C, Radtke T. The 1-Minute Sit-to-Stand Test in Lung Transplant Candidates: An Alternative to the 6-Minute Walk Test. Respir Care. 2020 Apr;65(4):437-443. doi: 10.4187/respcare.07124. Epub 2019 Oct 22. PMID 31641072
- [Background] Chhajed BS. Correlation between 6MWT, 2MST and TUG among Hypertensive Older Individuals.
- [Background] Nogueira MA, Almeida TDN, Andrade GS, Ribeiro AS, Rego AS, Dias RDS, Ferreira PR, Penha LRLN, Pires FO, Dibai-Filho AV, Bassi-Dibai D. Reliability and Accuracy of 2-Minute Step Test in Active and Sedentary Lean Adults. J Manipulative Physiol Ther. 2021 Feb;44(2):120-127. doi: 10.1016/j.jmpt.2020.07.013. Epub 2021 Jan 9. PMID 33431278
- [Background] Braghieri HA, Kanegusuku H, Corso SD, Cucato GG, Monteiro F, Wolosker N, Correia MA, Ritti-Dias RM. Validity and reliability of 2-min step test in patients with symptomatic peripheral artery disease. J Vasc Nurs. 2021 Jun;39(2):33-38. doi: 10.1016/j.jvn.2021.02.004. Epub 2021 Mar 19. PMID 34120695
- [Background] Bennett H, Parfitt G, Davison K, Eston R. Validity of Submaximal Step Tests to Estimate Maximal Oxygen Uptake in Healthy Adults. Sports Med. 2016 May;46(5):737-50. doi: 10.1007/s40279-015-0445-1. PMID 26670455